CLINICAL TRIAL: NCT06105450
Title: Potential Role of Diaphragmatic Muscle Weakness as a Cause of Persistent Exertional Dyspnea in Patients With COVID-19 Disease Without Hospitalization
Brief Title: Respiratory Muscle Assesment in COVID-patients Without Hospitalization
Acronym: RMA-COVID-19
Status: Completed | Type: Observational
Sponsor: RWTH Aachen University (Other)
Responsible Party: Principal Investigator, Jens Spießhöfer, Principal Investigator, RWTH Aachen University
Other Study IDs: 23-296
Record Dates: First submitted 2023-10-26; First posted 2023-10-27 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Covid19; Diaphragm Injury
Keywords: Respiratory muscle functtion
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples obtained based on venous puncture
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Comprehensive assessment of respiratory muscle function. — Comprehensive assessment of respiratory muscle function to the point of its invasive assessment with recordings of twitch transdiaphragmatic pressure in response to magnetic phrenic nerve stimulation and stimulation of the lower thoracic nerve roots.

SUMMARY:
Fatigue and exercise intolerance after survived COVID-19-infection might be related to weakness of the respiratory muscles. The aim of the project is to measure respiratory muscle function and strength in our respiratory physiology laboratory in patients who were not hospitalized during the acute COVID-19-infection but still complain of different persistent symptoms including exertional dyspnea and fatigue.

DETAILED DESCRIPTION:
Since the beginning of the COVID pandemic, more and more recovered patients have a number of persistent symptoms including exertional dyspnea and fatigue even months after recovering from acute coronavirus disease 2019 (COVID-19). These symptoms often cannot be explained because routine clinical diagnoses, including extensive cardiac and pulmonary examinations, do not reveal any relevant abnormalities.

In our previous study (Regmi et al) with 50 patients formerly hospitalized due to acute COVID-19 infection, it was shown that diaphragm muscle weakness contributes to persistent exertional dyspnea about one year after hospitalization for COVID-19, regardless of mechanical ventilation. Additionally, the severity of exertional dyspnea correlated with the extent of diaphragmatic weakness.

Since laboratory findings, pulmonary function tests and cardiological routine examinations did not reveal any significant impairments, this was the first time that a potential pathophysiological correlate is objectively associated with dyspnea in long COVID-19 syndrome. The results of our study were clinically relevant because the persistent symptom burden in patients after surviving COVID-19 infection remains very high. In addition diaphragm training presents itself as a potential therapeutic target, since in other diseases such as COPD, such training has been shown to improve the symptoms. Therefore, the investigators believe that the results provide important perspectives, both for the pathophysiological understanding and for the potential treatment of persistent exertional dyspnea in patients.

However, a considerable gap exists here: a significant number of patients who suffer from an acute COVID-19 infection but do not have a severe course during the initial infection, so that hospitalization is not necessary, still complain of different persistent symptoms. Here, too, despite an extensive cardiopulmonary work-up, there is a lack of a sufficient explanation of the lasting complaints. It is precisely in these patients that a possible role of diaphragmatic weakness on the symptoms is yet to be investigated using already established gold standard techniques.

ELIGIBILITY:
Inclusion Criteria:

* Patients with COVID-19 infection without hospitalization during the acute infection (n=25)
* Patients aged at least 18 years, who are mentally and physically able to consent and participate into the study

Exclusion Criteria:

* Clinically pre-established cardiovascular disease or other pulmonary diseases which might lead to exertional dyspnea (systolic heart failure, COPD).
* Body-mass-index (BMI) >40
* Expected absence of active participation of the patient in study-related measurements
* Alcohol or drug abuse
* Metal implant in the body that is not MRI compatible (NON MRI compatible pacemaker, implantable defibrillator, cervical implants, e.g. brain pacemakers etc.)
* Slipped disc
* Epilepsy
* Bound to a wheel chair

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 25 patients will be enrolled. Patients from the outpatient clinic of Department of Pneumology and Intensive Care UKA Aachen with a COVID infection at least six months ago without the need for hospitalization during the initial infection phase. Those patients will be compared with healthy controls (availaible data from pre-covid era) matched in a 3:1 ratio for age, sex and body mass index (BMI).
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Twitch transdiaphragmatic pressure in response to supramaximal magnetic stimulation of the phrenic nerve roots | 1 year
  Recording of twitch transdiaphragmatic pressure (Unit: Pressure in cmH2O)
Respiratory mouth pressures | 1 year
  Measurement of respiratory (inspiratory and expiratory) mouth pressures (Unit: Pressure in cmH2O)

SECONDARY OUTCOMES:
Diaphragm ultrasound | 1 year
  Comprehensive evaluation of diaphragm excursion (amplitude during tidal breathing, sniff maneuver and maximal inspiration in cm, corresponding velocity in cm/sec, respectively) and thickening on ultrasound (thickness at functional residual capacity, at total lung capactiy in cm), Markers of Diaphragm excursion and thickening will be combined to classify diaphragm function as normal, mildly, moderately or severly impaired.
Exercise intolerance | 1 year
  Comprehensive evaluation of symptoms (breathlesness based on NYHA class, on a visual scale ranging from 1-10, respectively) and exercise capacity (6 minute walking distance). These measurements will be combined to classifiy patients as presenting with exercise intolerance or no exercise intolerance.
Lung function | 1 year
  Comprehensive assessment of lung function by bodyplethysmography (most importantly forced vital capacity, forced expiratory volume after 1 second, intrathoracic gas volume, residual volume) and capillary blood gas analysis (most importantly pO2 in mmHG and pCO2 in mmHG). These measurements will be combined to classify patients as showing normal, restrictive, obstructive lung function impairment, as being hypoxic, hypercapnic, respectively.
EMG | 1 year
  Diaphragm and accessory respiratory muscle electromyography

CONTACTS AND LOCATIONS:
Overall Officials: Michael Dreher, Professor, Study Director — RWTH Aachen University; Jens Spiesshoefer, MD, Principal Investigator — RWTH Aachen University; Binaya Regmi, MD, Study Chair — RWTH Aachen University
Locations (1):
- Jens Spiesshoefer, Aachen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Regmi B, Friedrich J, Jorn B, Senol M, Giannoni A, Boentert M, Daher A, Dreher M, Spiesshoefer J. Diaphragm Muscle Weakness Might Explain Exertional Dyspnea 15 Months after Hospitalization for COVID-19. Am J Respir Crit Care Med. 2023 Apr 15;207(8):1012-1021. doi: 10.1164/rccm.202206-1243OC. PMID 36596223
- [Background] Spiesshoefer J, Herkenrath S, Henke C, Langenbruch L, Schneppe M, Randerath W, Young P, Brix T, Boentert M. Evaluation of Respiratory Muscle Strength and Diaphragm Ultrasound: Normative Values, Theoretical Considerations, and Practical Recommendations. Respiration. 2020;99(5):369-381. doi: 10.1159/000506016. Epub 2020 May 12. PMID 32396905
- [Background] Sudre CH, Murray B, Varsavsky T, Graham MS, Penfold RS, Bowyer RC, Pujol JC, Klaser K, Antonelli M, Canas LS, Molteni E, Modat M, Jorge Cardoso M, May A, Ganesh S, Davies R, Nguyen LH, Drew DA, Astley CM, Joshi AD, Merino J, Tsereteli N, Fall T, Gomez MF, Duncan EL, Menni C, Williams FMK, Franks PW, Chan AT, Wolf J, Ourselin S, Spector T, Steves CJ. Attributes and predictors of long COVID. Nat Med. 2021 Apr;27(4):626-631. doi: 10.1038/s41591-021-01292-y. Epub 2021 Mar 10. PMID 33692530
- [Background] Langer D, Ciavaglia C, Faisal A, Webb KA, Neder JA, Gosselink R, Dacha S, Topalovic M, Ivanova A, O'Donnell DE. Inspiratory muscle training reduces diaphragm activation and dyspnea during exercise in COPD. J Appl Physiol (1985). 2018 Aug 1;125(2):381-392. doi: 10.1152/japplphysiol.01078.2017. Epub 2018 Mar 15. PMID 29543134
- [Background] Griffin L, Cafarelli E. Resistance training: cortical, spinal, and motor unit adaptations. Can J Appl Physiol. 2005 Jun;30(3):328-40. doi: 10.1139/h05-125. PMID 16129897